CLINICAL TRIAL: NCT06592235
Title: Assessment of Awareness of Individuals with Chronic Lung Disease on Climate Change, Heat Waves, Air Pollution, and Their Interactions with Physical Activity
Brief Title: Awareness of Individuals with Chronic Lung Disease About Climate Change, Heat Waves, Air Pollution and Physical Activity
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Principal Investigator, Hacettepe University
Other Study IDs: SBA 24/794
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Climate Change; Chronic Lung Disease; Air Pollution

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Individuals with chronic obstructive lung disease: Individuals with chronic obstructive lung disease
  Interventions: Other: No intervention
- Individuals with asthma: Individuals with asthma
  Interventions: Other: No intervention
- Individuals with bronchiectasis: Individuals with bronchiectasis
  Interventions: Other: No intervention
- Individuals with interstitial lung disease: Individuals with interstitial lung disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Climate change is characterized by global temperature increase, melting of glaciers and increasing temperature of ocean waters. Increase in greenhouse gases such as nitrogen and carbon dioxide negatively affects air and water quality. Extreme events such as extreme heat waves, floods and hurricanes are events seen with climate change. It is known that climate change and air pollution have negative effects on public health. Its adverse effects are often seen in individuals with rhinosinusitis, asthma and chronic obstructive pulmonary disease. Air pollution is expected to increase due to the ongoing economic growth and population growth worldwide, resulting in more respiratory diseases and disease burden. This study aims to assess the awareness level of individuals with chronic lung disease on climate change, heat waves, air pollution and their interaction with physical activity and anxiety and depression levels, and to better understand the experiences of patients and learn their perspectives. Within the scope of the study, it is planned to provide patients brief information on this subject and receive feedback about this information.

ELIGIBILITY:
Inclusion criteria for the study:

* Being 18 years of age or older,
* Having a chronic lung disease (COPD, asthma, bronchiectasis, cystic fibrosis, interstitial lung disease) and being referred to the Cardiopulmonary Rehabilitation Unit of Hacettepe University, Faculty of Physical Therapy and Rehabilitation for cardiopulmonary physiotherapy and rehabilitation,
* Being clinically stable,
* Using a smartphone with a pedometer,
* To cooperate with the tests to be conducted,
* Being willing to participate in the study.

Exclusion criteria:

* Having had an acute exacerbation or having changed medication in the last month,
* Having a severe cardiovascular, orthopedic or neurological problem that may affect the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having a chronic lung disease (COPD, asthma, bronchiectasis, cystic fibrosis, interstitial lung disease)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Air temperature | 1 week before other assessments
  The air temperature of the province and district where the patients were located and lived one week before the assessment will be recorded from the open access website of the General Directorate of Meteorology of the Ministry of Environment and Urbanization (https://www.mgm.gov.tr/).
Humidity level | 1 week before other assessments
  The humidity level of the province and district where the patients were located and lived one week before the assessment will be recorded from the open access website of the General Directorate of Meteorology of the Ministry of Environment and Urbanization (https://www.mgm.gov.tr/).
Wind speed | 1 week before other assessments
  The wind speed of the province and district where the patients were located and lived one week before the assessment will be recorded from the open access website of the General Directorate of Meteorology of the Ministry of Environment and Urbanization (https://www.mgm.gov.tr/).
Air pollution | 1st day
  The province and district where the patients were located and lived in the last week before the assessment will be recorded and the air pollutant values of PM2.5, PM10, CO, NO2, SO2, NO, O3 in the settlement where they lived in the last week will be accessed from the open access website of the continuous monitoring center of the Ministry of Environment and Urbanization and will be recorded and used for analysis. (https://sim.csb.gov.tr/STN/STN_Report/StationDataDownloadNew).
Cognitive assessment | 1st day
  Standardized Mini Mental Test. will be used for cognitive assessment. It provides assessment of cognitive activities such as understanding, reading, remembering and performing actions consisting of eleven questions. It is scored between 0-30. &amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;lt; 18 (quite a lot of cognitive impairment), 18-22 (moderate cognitive impairment), 23-26 (low cognitive impairment), 27-30 (no cognitive impairment).
Anxiety and depression assessment | 1st day
  Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety and depression. Seven out of a total of 14 questions measure anxiety and seven questions assess depression. The answers are scored in a four-point Likert format and between 0 and 3. The lowest score that patients can get from both subscales is 0, and the highest score is 21.
Assessment of quality of life | 1st day
  The St. George Respiratory Questionnaire (SGRQ) will be used to assess disease-specific quality of life. The SGRQ is a questionnaire consisting of three categories that patients answer themselves, assessing symptoms, activities and the impact of their disease on their daily lives. The questionnaire consists of a total of 76 questions and is scored between zero and 100, with high scores indicating poor health status.
Health literacy assessment | 1st day
  The Rapid Assessment of Adult Health Literacy in Medicine (REALM) scale will be used for health literacy assessment. REALM tests people&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s word recognition and pronunciation skills. It is a word recognition test in which 66 health-related words are given, with the words becoming increasingly more difficult. Patients will be asked to read all of these words out loud in order.
Physical activity assessment | 1st day
  Physical activity level will be assessed using the International Physical Activity Questionnaire (IPAQ) (Short Form). This questionnaire was designed as a short and long form to determine the physical activity and sedentary behavior levels of adults. The IPAQ short form consists of seven questions and provides information on the time spent in vigorous activity, moderate activity and walking activities, as well as the time spent sitting. Higher IPAQ scores reflect greater levels of physical activity. In addition, the step counts of the participants for the last week will be recorded from their smartphones.

SECONDARY OUTCOMES:
Respiratory functions | 1st day
  Respiratory function test values will be recorded from patient records.
Body mass index | 1st day
  Body mass index value will be calculated.
Disease-related symptoms | 1st day
  Disease-related symptoms (shortness of breath, cough and sputum) will be questioned and recorded.
Socio-economic status | 1st day
  Socio-economic status will be recorded.
Education level | 1st day
  Education level will be recorded.
Dyspnea assessment | 1st day
  Modified Medical Research Council (mMRC) dyspnea scale will be used for dyspnea assessment. mMRC dyspnea scale is a scale in which individuals choose the expression that best describes their dyspnea levels from five expressions related to shortness of breath. It easily evaluates shortness of breath due to its simplicity and reliability. Higher mMRC dyspnea scale scores indicate more severe dyspnea (breathlessness).
Charlson Comorbidity Index | 1st day
  Charlson Comorbidity Index (CCI) will be used to query accompanying comorbidities. Higher CCI scores indicate a greater burden of comorbid conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Aslihan Cakmak-Onal, PhD, PT, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, PT, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Amato G, Cecchi L, D'Amato M, Annesi-Maesano I. Climate change and respiratory diseases. Eur Respir Rev. 2014 Jun;23(132):161-9. doi: 10.1183/09059180.00001714. No abstract available. PMID 24881071
- [Background] Ebi KL, Vanos J, Baldwin JW, Bell JE, Hondula DM, Errett NA, Hayes K, Reid CE, Saha S, Spector J, Berry P. Extreme Weather and Climate Change: Population Health and Health System Implications. Annu Rev Public Health. 2021 Apr 1;42:293-315. doi: 10.1146/annurev-publhealth-012420-105026. Epub 2021 Jan 6. PMID 33406378
- [Background] Tran HM, Tsai FJ, Lee YL, Chang JH, Chang LT, Chang TY, Chung KF, Kuo HP, Lee KY, Chuang KJ, Chuang HC. The impact of air pollution on respiratory diseases in an era of climate change: A review of the current evidence. Sci Total Environ. 2023 Nov 10;898:166340. doi: 10.1016/j.scitotenv.2023.166340. Epub 2023 Aug 15. PMID 37591374
- [Background] Eguiluz-Gracia I, Mathioudakis AG, Bartel S, Vijverberg SJH, Fuertes E, Comberiati P, Cai YS, Tomazic PV, Diamant Z, Vestbo J, Galan C, Hoffmann B. The need for clean air: The way air pollution and climate change affect allergic rhinitis and asthma. Allergy. 2020 Sep;75(9):2170-2184. doi: 10.1111/all.14177. Epub 2020 Jan 30. PMID 31916265
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716